CLINICAL TRIAL: NCT01305343
Title: Evaluation of Neurologic Complications Associated With Surgical Correction of Adult Spinal Deformity: A Prospective, Observational, Multi-center Study
Brief Title: Neurologic Complications in Spinal Deformity Surgery
Status: Completed | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Collaborators: Scoliosis Research Society (Other)
Responsible Party: Sponsor
Other Study IDs: Scoli-Risk-1
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Adult Spinal Deformity
Keywords: Spinal Deformity; Scoliosis; Neurologic complications
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgical treatment: This observational study is examining the outcomes of standard surgical treatments for adult spinal deformity.
  Interventions: Procedure: Routinely performed surgical correction of spinal deformity

INTERVENTIONS:
Procedure: Routinely performed surgical correction of spinal deformity — Routinely performed surgical correction of spinal deformity

SUMMARY:
240 subjects with "high risk" adult spinal deformity requiring surgical correction will be enrolled in a prospective multi-center international study. "High risk" patients are defined by either their diagnoses and/or the type of surgical intervention as listed in the inclusion criteria. Neurologic complications in the form of new motor and sensory deficits will be monitored prospectively in all patients at hospital discharge, and at 6 weeks (± 2 weeks) six months (± 2 months) and 24 months(± 2 months) after the surgery. All new deficits will be adjudicated for relationship to the surgical intervention.

Regression analyses will be used to evaluate the association between patient demographics, co morbidities, treatment history, spinal deformity characteristics, surgical characteristics, non-neurologic complications and pre-surgical status to occurrence of a neurologic deficit after surgery.

DETAILED DESCRIPTION:
Although the incidence of complications in patients undergoing correction of their spinal deformity has been reported extensively, the majority of these studies were retrospective. There were only five studies, three from a single institution, with prospectively collected data that specifically identified complications. The largest series was from Buchowski et al who reported on 108 patients with fixed sagittal deformity undergoing Pedicle Subtraction Osteotomy (PSO) with a 14% over-all complication rate with motor weakness in 11 patients and neurogenic bladder in one patient, of which 3 were permanent. Yang reported on 35 patients undergoing PSOs with a 46% over-all complication rate and one transient nerve root motor deficit. Ahn in 2002 reported on 83 patients undergoing various osteotomies for sagittal imbalance and reported a 34% over-all complication rate with 3 permanent and 3 transient nerve root deficits.

Given this lack of information, there is a need to determine the true incidence of complications using a prospective multi-center design. There is a need to identify neurologic deficits in a more systematic fashion to include spinal cord, cauda equina and nerve root deficits as well as radiculopathies. The risk factors associated with the occurrence of a complication, especially a neurologic complication, also needs to be more fully elucidated. This is increasingly relevant, as newer surgical techniques allow for more aggressive correction of the spinal deformity that may put the spinal cord and nerve roots at increased risk. Valid data on the incidence and types of neurologic deficits is also needed in order to study newer drugs that are available that may mitigate this risk.

The primary objectives of this study are: (i) to establish the incidence of neurologic deficit in "high risk" adult patients undergoing correction of their spinal deformity of adult spinal deformity and (ii) to identify characteristics associated with increased risk of neurologic complications. Secondary objectives include (i) to determine the incidence of all complications related to surgical correction of "high risk" adult spinal deformity; (ii) to determine the short-term clinical outcomes in patients undergoing correction of their spinal deformity and (iii).to determine amount of radiographic and clinical correction of deformity

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 to 80 years old inclusive
* Diagnosis of adult spinal deformity with an apex of the major deformity in the cervico-thoracic or thoraco-lumbar region (Apex between C7 and L2 inclusive) with any of the following deformity characteristics

  * Primary Scoliosis, Kyphosis or Kyphoscoliosis with major Cobb ≥ 80° in the coronal or sagittal plane
  * Congenital Spinal Deformity undergoing corrective spinal osteotomy
  * Revision Spinal Deformity undergoing corrective spinal osteotomy
* Any patient undergoing a 3-column spinal osteotomy (i.e. Pedicle Subtraction Osteotomy, Vertebral Column Resection) from C7 to L5 inclusive
* Any patient with preoperative myelopathy due to their spinal deformity
* Any patient with ossification of the Ligamentum Flavum or Posterior Longitudinal Ligament and a deformity that needs concomitant reconstruction along with decompression of the spinal cord

Exclusion Criteria:

* Unlikely to comply with follow-up
* Recent history ≤ 3 months of substance dependency or psychosocial disturbance
* Presence of active malignancy
* Has active, overt bacterial infection, systemic or local
* Recent (≤3 months) history of significant spinal trauma/injury/ fracture/malignancy in the spinal region
* Patients with complete, long term paraplegia
* Pregnant or nursing women, unable to agree not to become pregnant for a period of 6 months after surgery
* Prisoners
* Institutionalized individuals

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving care at the investigative sites will be pre-screened as potential subjects for this observational study study.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Rate of treatment-related neurologic complication | 6 months
  * Spinal Cord Deficit
  * Cauda Equina Deficit
  * Nerve Root Deficit
    * Motor Deficit
    * Sensory Deficit
    * Radiculopathy

SECONDARY OUTCOMES:
• Sensory status as measured by the ASIA Sensory Score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lenke, MD, Principal Investigator — Scoliosis Research Society
Locations (15):
- United States (8):
  - University of California, San Francisco, California
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Department of Orthopaedic Surgery, Washington University School of Medicine, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - NYU School of Medicine, Yew York, New York
  - University of Virginia, Charlottesville, Virginia
- University of Toronto, Toronto, Canada
- China (2):
  - University of Hong Kong, Hong Kong
  - Nanjing Drum Tower Hospital, Nanjing
- Rigshospitalet, Copenhagen, Denmark
- University School of Medicine, Hamamatsu, Japan
- Hospital Universitari Vall D'Hebron, Barcelona, Spain
- University Hospital Nottingham, NHS Trust, Nottingham, United Kingdom

REFERENCES:
- [Derived] Kwan KYH, Lenke LG, Shaffrey CI, Carreon LY, Dahl BT, Fehlings MG, Ames CP, Boachie-Adjei O, Dekutoski MB, Kebaish KM, Lewis SJ, Matsuyama Y, Mehdian H, Qiu Y, Schwab FJ, Cheung KMC; AO Spine Knowledge Forum Deformity. Are Higher Global Alignment and Proportion Scores Associated With Increased Risks of Mechanical Complications After Adult Spinal Deformity Surgery? An External Validation. Clin Orthop Relat Res. 2021 Feb 1;479(2):312-320. doi: 10.1097/CORR.0000000000001521. PMID 33079774
- See also: Related Info — http://www.aospine.org
- See also: Related Info — http://www.srs.org/